CLINICAL TRIAL: NCT04478721
Title: Randomised Controlled Trial of Temocillin vs Meropenem for the Targeted Treatment of Bacteraemia Due to Enterobacteriaceae Showing Resistance to Third Generation Cephalosporins
Brief Title: Temocillin vs Meropenem for the Targeted Treatment of Bacteraemia Resistant to Third Gen Cephalosporins
Acronym: ASTARTÉ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other); Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASTARTÉ; 2020-000064-39 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-07-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bacteremia
Keywords: Bacteraemia; Enterobacteriaceae; Temocillin; Third-generation cephalosporin-resistant Enterobacteriaceae.
MeSH Terms: conditions — Bacteremia; Toxemia | interventions — temocillin; Meropenem

STUDY DESIGN:
Intervention Model Description: Randomized 1.1 to temocillin: meropenem
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temocillin (Experimental): Patients enrolled in this arm, will receive 2g each 8 hours of intravenous temocillin.
  Interventions: Drug: Temocillin
- Meropenem (Active Comparator): Patients enrolled in this arm, will receive 1g each 8 hours of intravenous meropenem.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Temocillin — The intervention of experimental arm will be Intravenous administration of temocillin.
  Arms: Temocillin
Drug: Meropenem — The intervention of comparator arm will be intravenous administration of meropenem.
  Arms: Meropenem

SUMMARY:
A Phase 3, Multicenter, Randomised, Controlled, Open-Label Study to demonstrate noninferiority of temocillin (unauthorized investigational medicinal product IMP in Spain, but authorized in Belgium and UK) vs a carbapenem antibiotic (meropenem) in adults with bacteraemia due to third-generation cephalosporin-resistant Enterobacteriaceae.

The duration of treatment will be between 7 and 14 days. From the 5th day of intravenous treatment, the sequential oral treatment is permitted if the patient meets appropriate conditions.

DETAILED DESCRIPTION:
The objective of the trial is to demonstrate the non-inferiority of temocillin (2g each 8 hours, intravenous) to carbapenems (meropenem 1g each 8 hours, intravenous) in terms of efficacy and safety in the targeted treatment of bacteraemia due to Enterobacteriaceae resistant to third-generation cephalosporins, and therefore provide evidence for the use of temocillin in these infections.

The duration of treatment will be between 7 and 14 days. From the 5th day of intravenous treatment, the sequential oral treatment is permitted if the patient meets appropriate conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with monomicrobial bacteremia due to Enterobacteriaceae showing resistance to cefotaxime, ceftriaxone (MIC >2 mg/L) and/or ceftazidime (MIC >4 mg/L), and sensible to temocillin (MIC ≤8 mg/L, except in bacteremia only of urinary origin, for which the criterion is MIC ≤16 mg/L ) and meropenem (MIC ≤2 mg/L).

Patients with polymicrobial bacteremia caused by more than one Enterobacteriaceae species may also be included, provided at least one of them is resistant to third-generation cephalosporins, and both are susceptible to meropenem and temocillin.

* Duration of intravenous treatment is planned to be at least 4 days from randomization, or 3 days if the empirical treatment prior to randomization was active.
* The patient signed informed consent form.
* Potentially fertile patients must have a negative pregnancy test.

Exclusion Criteria:

* <18 years
* Pregnancy
* Breastfeeding
* Terminal condition, with life expectancy of less than 30 days, or palliative care , such that no actions will be taken to control the source of infection if necessary. Patients receiving palliative care with a life expectancy greater than 30 days may be included if source control is not necessary or, if necessary, will be carried out.
* Allergy to betalactams
* Polymicrobial bacteraemia (except when the other microorganism is considered a contaminant, (e.g. coagulase-negative staphylococci or diphtheroids in a single blood culture, or in cases where more than one Enterobacteriaceae species is isolated, provided that at least one isolate is resistant to third-generation cephalosporins and both are susceptible to meropenem and temocillin).
* Infections typically needing prolonged >14 days of therapy (e.g., endocarditis, prosthetic joint infection, vascular graft infection, empyema, chronic prostatitis) or meningitis. Patients who initially do not have a confirmed diagnosis of these infections may be included; if the diagnosis is made subsequently, the patient may be kept in the trial at the discretion of the investigator, establishing the duration of treatment that he considers necessary.
* Active empirical treatment> 96 hours after initial blood culture extraction
* Delay in inclusion> 48 h
* Recruited in another clinical trial with active treatment
* Peritoneal dialysis or continuous hemofiltration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with a "success" at the test of cure (TOC) | Up to 7-10 days after the last day of antibiotic therapy
  A success at the test of cure is the resolution of infection symptoms
Survival at day 28 | At day 28.
  Number of patients who are alive
Number of patients who do not need to stop or change the assigned drug | Up to 7-14 days after the last day of antibiotic therapy
  Reasons for not change can be no adverse event, no perceived failure during treatment or no occurrence of a superimposed infection.
  Participants who stop or change the assigned drug will not meet the primary outcome.
Number of patients who do not need to prolong therapy beyond 14 days | Up to 7-14 days after the last day of antibiotic therapy
  Assigned treatment to be administered for less than 14 days
Not recurrence until day 28 | At day 28.
  Recurrence is reappearance of symptoms with positive blood culture for the same microorganism.
  Participants with recurrence will not meet the primary outcome.

SECONDARY OUTCOMES:
28-day mortality | Up to day 28.
  Number of patients dead up to day 28.
Length of hospital stay (days) | Through study completion, an average of 28 days
  Number of days patients has been in-hospital
Length of intravenous therapy (days) | From day 1 of intravenous antibiotic treatment administration to last intravenous administration, average 14 days
  Number of days patients has been under intravenous antibiotic treatment
Length of total administration of therapy (days) | From day 1 of intravenous or oral antibiotic treatment administration to last intravenous or oral administration, average 14 days
  Number of days patients has been under intravenous or oral antibiotic treatment
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to day 28
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Number of subjects with resistance development during therapy | Up to day 28
  Resistance development will be measured in a positive blood culture
Recurrence rate | Up to day 28.
  Percentage of subjects with recurrence
Changes in Sequential Organ failure (SOFA) score | At days 1, 3, end of treatment (days 7-14) and visit 4
  Sequential Organ failure (SOFA) score changes
Changes in Barthel Index for Activities of Daily Living (ADL) for patients older than 70 years old | At days 1, 3, end of treatment (days 7-14) and visit 4
  Barthel Index for Activities of Daily Living (ADL) score changes; score from 0, completely dependent patient to 100, completely independent for activities of daily living
Number of subjects with development of superimposed infections. | Up to day 28.
  Development of superimposed infections will be measured in a positive culture

OTHER OUTCOMES:
Peak Plasma Concentration (Cmax) of temocillin | At 1hour, 4hours, 6hours and y 8hours from temocillin first infusion, on days 1 and 3
  Exploratory objective in a reduced number of patients on which plasma levels of temocillin will be measured to determine maximum plasma levels of temocillin
Minimum Plasma Concentration (Cmin) of temocillin | At 1hour, 4hours, 6hours and y 8hours from temocillin first infusion, on days 1 and 3
  Exploratory objective in a reduced number of patients on which plasma levels of temocillin will be measured to determine minimum plasma levels of temocillin
Area under the plasma concentration versus time curve (AUC) of temocillin | At 1hour, 4hours, 6hours and y 8hours from temocillin first infusion, on days 1 and 3
  Exploratory objective in a reduced number of patients on which plasma levels of temocillin will be measured to determine area under curve of temocillin

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodriguez Baño, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (29):
- Spain (29):
  - Hospital ParcTaulí, Sabadell, Barcelona
  - Hospital Universitario Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario de Puerto Real, Puerto Real, Cádiz
  - Complejo Hospitalario San Millán-San Pedro De La Rioja, Logroño, La Rioja
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Complejo Hospitalario Universitario La Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Locus Augusti, Lugo, Lugo
  - Hospital Universitario de la Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitari Son Espases, Palma
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Complejo Hospitalario Universitario de Vigo, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Planning for the study will be shared with potential sites pertaining to Spanish Network for Research in Infectious Disease (REIPI)for participation. IPD is not foreseen out of this groups due to the specific characteristics of patients and sites to be candidates for study participation.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: From starting to three years of study completion planification
Access Criteria: Spanish Network for Research in Infectious Disease investigators

REFERENCES:
- [Derived] Marin-Candon A, Rosso-Fernandez CM, Bustos de Godoy N, Lopez-Cerero L, Gutierrez-Gutierrez B, Lopez-Cortes LE, Barrera Pulido L, Borreguero Borreguero I, Leon MJ, Merino V, Camean-Fernandez M, Retamar P, Salamanca E, Pascual A, Rodriguez-Bano J; ASTARTE Study Group. Temocillin versus meropenem for the targeted treatment of bacteraemia due to third-generation cephalosporin-resistant Enterobacterales (ASTARTE): protocol for a randomised, pragmatic trial. BMJ Open. 2021 Sep 27;11(9):e049481. doi: 10.1136/bmjopen-2021-049481. PMID 34580096

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-04-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT04478721/SAP_000.pdf